CLINICAL TRIAL: NCT05707975
Title: Eco-anxiety and Severity of Suicide Risk in Adolescents
Brief Title: Eco-anxiety and Suicide
Acronym: EcoAnx
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_1118
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Suicide; Suicide Attempt; Suicidal; Anxiety
Keywords: Suicide risk; Eco-Anxiety; Adolescents
MeSH Terms: conditions — Suicide; Suicide, Attempted; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adolescents hospitalized in the service: Adolescents between 12 and 16 years old Intervention: filling of three scales (CAS, C-SSRS, HAD)
  Interventions: Other: Identifying a relationship between the intensity of eco-anxiety and the severity of suicide risk in adolescents

INTERVENTIONS:
Other: Identifying a relationship between the intensity of eco-anxiety and the severity of suicide risk in adolescents — Relationship between the intensity of eco-anxiety with the 13-item CAS score, and the seriousness of the suicide risk with the C-SSRS score

SUMMARY:
Suicide is a major public health problem. About 9,000 suicides per year are retrieved by year in France. Between 15,000 and 20,0000 suicide attempts give rise to contact with the healthcare system.

Among young people aged 15 to 24 years old, suicide is the second main cause of death. In this way, suicide among adolescents is a major public health priority, due to its seriousness, its frequency, and its potentially preventable nature.

The severity of suicide risk can be assessed by different scales, and the Columbia-Suicide Severity Rating Scale (C-SSRS) is the most widely used in the international literature for adolescents, assessing four dimensions: suicidal ideation, severity of ideation, suicidal behavior and lethality. The measurement of the seriousness of the suicide risk is therefore defined as the measurement of the importance of the direct and indirect negative consequences associated with this risk. It can be catch up in the four factors mentioned above.

Anxiety is one of the central pillars influencing the suicidal risk of adolescents. Very few studies have identified operationalizable and generalizable risk factors for anxiety. However, in adolescents, one of the risk factors for anxiety seems particularly important, because it is a factor that is both generic (i.e., it can be found in different profiles of adolescents), related to the projection in the future (which characterizes this population), and relatively specific to this age group, while being operational through validated questionnaires. This important risk factor is the eco-anxiety, which corresponds to anxiety related to climate change.

The theme of climate change is certainly a central social issue, but also an important public health issue. First, climate change raises direct risks to human health, and indirectly some risks for mental health. For instance, the direct consequences of a drought or natural disaster can cause material hardship that impacts indirectly mental health (Thoma et al., 2021). Secondly, climate change can also raise direct risk for mental health, and especially the eco-anxiety which is not the consequence of a direct risk from the environment on an individual, but rather constitutes mental distress related to the fear of such changes.

Eco-anxiety can be identified and measured in a valid and reliable way thanks to a scale used in the international literature, the "Climate Anxiety Scale" (CAS), which was validated in 2020 with 22 items with 4 factors by Clayton and Karazsia (Clayton and Karazsia, 2020), and translated and validated in French in 2022 by Mouguiama-Daouda (Mouguiama-Daouda et al., 2022), retaining as the most appropriate model the version with the first 13 items. This scale is suitable for adolescents from the age of 12 years old.

This 13-item scale is composed of two subscales that assess cognitive and emotional difficulties in response to climate change and functional impairment. Two subscales are added to this 13-item scale (and thus are part of the 22-item CAS also validated), which assess 1) direct or indirect personal experience of climate change, and 2) behavioral commitment and the tendency to deploy adaptive behavioral responses to climate change.

The literature reports a correlation between eco-anxiety and depression (Mouguiama-Daouda et al., 2022). Indeed, depressive symptoms can influence how people worry about climate change. The correlation between eco-anxiety and anxiety is variable in the literature and has been studied using questionnaires focusing on generalized anxiety (Mouguiama-Daouda et al., 2022). Higher suicide rates have certainly been shown in populations affected by climate change (Dumont et al., 2020), related to the direct consequences of climate change, e.g., due to pollution, increased temperature or drought.

However, to the knowledge of the investigators and despite the major public health impact in adolescents, no study has investigated the relationships between eco-anxiety and the severity of suicide risk.

This study therefore seeks to examine the association between eco-anxiety in adolescents, assessed using the French version of the CAS, and the severity of suicide risk, assessed using the French version of the C-SSRS. We hypothesize that there would be a relationship between eco-anxiety and the severity of suicide risk in adolescents. Such results would allow both to refine the understanding of the risk of suicide, in its relationship with a central theme of society and public health, and to better identify and prevent behaviors at risk of suicide among adolescents.

ELIGIBILITY:
Inclusion Criteria:

- Adolescents aged 12 to 16, hospitalized at the Hopital Femme Mère Enfant, in the child and adolescent psychopathology department

Exclusion Criteria:

* Patient who does not speak French
* Patient unable to read or write.
* Patient with an intellectual development or oral comprehension disorder (eg severe dysphasia preventing understanding of the explanations given, or severe dyslexia preventing the reading of scale items).
* Oral or written refusal by the parents or the child.
* Child not affiliated to a social security system and under legal protection

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients hospitalized in the child and adolescent psychopathology department at the HFME
Sampling Method: Probability Sample
Enrollment: 261 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2026-10-27 (Estimated); Study Completion 2026-11-27 (Estimated)

PRIMARY OUTCOMES:
Relationship between the intensity of eco-anxiety with the 13-item CAS score, and the severity of suicide risk with the C-SSRS score | At the inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Femme Mère Enfant, Bron, Rhone, France

IPD SHARING:
Plan to Share IPD: No